CLINICAL TRIAL: NCT03391375
Title: An Open Label Phase I Clinical Trial to Evaluate the Effect of Late Boost on HIV-uninfected Vaccinees From EV06 Trial
Brief Title: Evaluation of the Effect of Late Boost on HIV-uninfected Vaccines From EV06 Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EuroVacc Foundation (Other)
Collaborators: MRC/UVRI and LSHTM Uganda Research Unit (Other); International AIDS Vaccine Initiative (Network); Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EV07
Record Dates: First submitted 2017-12-11; First posted 2018-01-05 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2017-12

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — AIDSVAX B-E

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DNA-Protein (Experimental): Co-administration of DNA-HIV-PT123 and AIDSVAX B/E at week 0, 4 and 24
  Interventions: Biological: DNA-HIV-PT123 & AIDSVAX B/E

INTERVENTIONS:
Biological: DNA-HIV-PT123 & AIDSVAX B/E — DNA-HIV-PT123 encodes clade C ZM96 Gag and gp140, CN54 Pol-Nef; AIDSVAX®B/E is a subtype B (MN) and subtype E (A244) HIV gp120 glycoprotein adsorbed onto aluminium hydroxide gel adjuvant

SUMMARY:
EV07 is an open label phase I clinical trial to evaluate the effect of late boost on HIV-uninfected vaccinees from EV06 trial.

The outcome of the EV06 trial has shown that the vaccine regimen is safe and well tolerated. Preliminary antibody immunogenicity analysis has demonstrated that the DNA/gp120 protein vaccine regimen induced strong gp120, gp140 and V1V2 region-focused binding IgG and neutralizing antibody responses. There is also preliminary evidence that S. mansoni infection may modulate antibody responses induced by vaccination1.

Based on these preliminary immunogenicity results of the EV06 study, a study with an additional boost with DNA-HIV-PT123 and AIDSVAX®B/E (Late Boost) is warranted in order to better investigate and understand the effects of the late boost on the response rate, magnitude and durability of vaccine induced immune responses.

The primary objective of EV07 is to evaluate the ability of the late boost combination of DNA-HIV-PT123 and AIDSVAX® B/E to enhance the pre-existing vaccine induced antibody responses.

ELIGIBILITY:
Inclusion Criteria:

1. Participated in the EV06 trial and received all three vaccinations from EV06 trial
2. HIV uninfected adults, as confirmed by a medical history, physical exam, and laboratory tests during screening
3. Able and willing to provide written informed consent prior to screening
4. Aged at least 18 at the time of consent
5. Able and willing to complete screening (about 1 month) and available for the planned follow-up period (6 months)
6. Willing to undergo HIV testing, risk reduction counselling and receive HIV test results
7. If female of childbearing potential (unless sterilised), willing to use a non-barrier contraceptive method from screening through the end of the study. Acceptable contraceptive methods include hormonal contraceptives (injection, transdermal patch, or implant) and intrauterine device (IUD).
8. If male, willing to use male condoms and not make a woman pregnant from enrolment through the end of the study.
9. Willing to provide blood, urine and stool samples for laboratory examination

Exclusion Criteria:

1. HIV-1/2 infection
2. Symptomatic and asymptomatic malaria infection (presence of malaria parasites on thick blood smear)
3. Clinically significant acute or chronic illness at the time of randomization.
4. Any clinically relevant abnormality on history or examination
5. Use of immunosuppressive medication (other than inhaled or topical immunosuppressants)
6. Receipt of immunoglobulin within past 60 days
7. Abnormal laboratory values as specified below from blood collected within 42 days prior to randomization:

   1. Hematology

      * Haemoglobin <9.0 g/dL or <5.59 mmol/L
      * Absolute Neutrophil Count (ANC): < 1000/mm3 or < 1.0 x 109/L
      * Absolute Lymphocyte Count (ALC): ≤ 500/mm3 or ≤ 0.5 x 109/L
      * Platelets: ≤ 90,000 ≥ 550,000/mm3 or ≤ 90 x 109 ≥ 550 x 109/L
   2. Chemistry

      * Creatinine: > 1. 1 x ULN
      * AST: >2.6 x ULN
      * ALT: >2.6 x ULN
   3. Urinalysis: abnormal dipstick confirmed by microscopy

      * Protein 2+ or more
      * Blood 2+ or more (not due to menses)
8. History or evidence of autoimmune disease.
9. Positive for Hepatitis B surface antigen (HbsAg), positive for antibodies to Hepatitis C virus (HCV) or active syphilis.
10. Receipt of blood or blood products within the previous 6 months
11. History of severe allergic reactions to any substance requiring hospitalization or emergency medical care (e.g. Steven-Johnson syndrome, bronchospasm or hypotension)
12. Prior or current participation in another investigational agent trial except to the EV06 trial
13. Current anti-tuberculosis (TB) prophylaxis or therapy
14. If female, currently pregnant (positive serum or urine pregnancy test), planning to get pregnant in the next 9 months or lactating
15. History or evidence of any systemic disease or any acute or chronic illness that, in the opinion of the investigator, may compromise the volunteer's safety or interfere with the evaluation of the safety or immunogenicity of the vaccine

Volunteers will be enrolled regardless of schistosomiasis infection status. Volunteers with high S. mansoni egg count of >2000 eggs per gram of stool at screening will be treated before vaccination. Volunteers with low S mansoni egg count of <2000 eggs per gram of stool at screening will be asked to forgo treatment until after completion of week 24 visit of the trial. Volunteers with other helminth infections at screening will also receive treatment before vaccination.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Vaccine induced binding antibody responses | week 24
  HIV-specific Env binding Antibody response
Vaccine induced neutralizing antibody responses | week 24
  Neutralizing antibody responses against tier 1 and tier 2 HIV-1 isolates
Safety and tolerability of the late boost vaccination | 7 days follow-up period after the late boost
  Proportion of volunteers with local and systemic reactogenicity events
Safety and tolerability of the late boost vaccination | 4-week follow-up period after the late boost
  Proportion of volunteers with adverse events
Safety and tolerability of the late boost | Up to 24 weeks
  Proportion of volunteers with serious adverse events

SECONDARY OUTCOMES:
Ability of the late boost combination of DNA-HIV-PT123 and AIDSVAX® B/E to enhance the pre-existing vaccine induced T-cell responses | Week 2, 12 and 24
  HIV-specific CD4 and CD8 T cell responses

CONTACTS AND LOCATIONS:
Overall Officials: Pontiano Kaleebu, Principal Investigator — MRC/UVRI and LSHTM Uganda Research Unit
Locations (1):
- Uganda Virus Research Institute - International AIDS Vaccine Initiative HIV Vaccine Program (UVRI-IAVI), Entebbe, Uganda

IPD SHARING:
Plan to Share IPD: No